CLINICAL TRIAL: NCT00481559
Title: An Open-Label Treatment Protocol for the Use of Voraxaze as Adjunctive Treatment for Patients Experiencing or at Risk of Methotrexate Toxicity
Brief Title: Treatment Protocol of Voraxaze for Patients Experiencing or at Risk of Methotrexate Toxicity
Status: Approved for marketing | Type: Expanded Access
Sponsor: BTG International Inc. (Other)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Other Study IDs: PR001-CLN-pro016
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Neoplasms
Keywords: Voraxaze; glucarpidase; carboxypeptidase; cancer; lymphoma; leukemia; osteosarcoma; methotrexate; delayed elimination; renal insufficiency; toxicity
MeSH Terms: conditions — Neoplasms; Lymphoma; Leukemia; Osteosarcoma; Renal Insufficiency | interventions — glucarpidase; Carboxypeptidases

INTERVENTIONS:
Drug: Voraxaze (glucarpidase) — 50 Units/kg in a bolus intravenous injection over 5 minutes
  Other Names: carboxypeptidase; CPG2; CPDG2

SUMMARY:
This protocol is for the treatment of toxic plasma methotrexate concentrations (>1 micromole per liter) in patients with delayed methotrexate clearance due to impaired renal function

DETAILED DESCRIPTION:
This treatment protocol will be available on a cost recovery basis to IRB-approved Investigators treating an eligible patient at any site in the US. In order to continue to make Voraxaze™ available following FDA approval and prior to being commercially available. Protherics needs to charge for the product, so there will be a cost to obtain Voraxaze™ under the Open-Label Treatment Protocol. Protherics is permitted under the FDA regulations (21 CFR 312.8) to charge for Voraxaze, to recover those costs associated with its manufacture, research and development, and handling, but do not include other commercial costs (profit).

Patient eligibility is based on MTX concentrations and laboratory values obtained per standard of care. Once an Investigator identifies a potential patient, he/she will contact the Voraxaze central call center (1-877-398-9829) to receive information regarding drug shipment. Eligible patients will have routine demographic, MTX, and Voraxaze therapy information collected.

Each patient will receive a single dose of Voraxaze 50 Units/kg in a bolus intravenous injection over 5 minutes. In addition to Voraxaze, patients will continue to receive standard of care treatment including leucovorin therapy, and supportive care such as hydration, alkalinization of urine and, if necessary, hemoperfusion/dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of any age who are experiencing delayed MTX clearance due to impaired renal function will be eligible to receive Voraxaze if the have toxic plasma MTX concentrations (>1 micromole per liter).

Exclusion Criteria:

* Voraxaze is not indicated for use in patients who exhibit the expected clearance of MTX (plasma MTX concentrations within 2 standard deviations of the mean MTX excretion curve specific for the dose of MTX administered) or those with normal or mildly impaired renal function because of the potential risk of sub therapeutic exposure to MTX.
* Patients with known hypersensitivity to Voraxaze (glucarpidase, carboxypeptidases)

Patients intolerant to lactose in food (e.g., dairy products) can still receive Voraxaze.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Paul Litka, MD, Study Chair — BTG (contract)